CLINICAL TRIAL: NCT03086057
Title: Optimizing Pre-exposure Prophylaxis (PrEP) Uptake & Adherence Among MSW Using a 2-stage Randomization Design
Brief Title: Optimizing PrEP Uptake & Adherence Among Male Sex Workers (MSW) Using a 2-stage Randomization Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Matthew Mimiaga, ScD, MPH, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R34MH110369-01 (NIH)
Record Dates: First submitted 2017-03-08; First posted 2017-03-22 (Actual); Results first posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-02

CONDITIONS: Prevention
Keywords: PrEP; Prevention; Male Sex Workers (MSW)
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Intervention Model Description: In Stage 1, individuals will be randomized (1:1) to receive the experimental PrEP navigation or standard of care. Among those who uptake PrEP in Stage 1, we will randomize those participants in Stage 2 (1:1) to receive the experimental adherence counseling or standard of care.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Strength Based Case Management (Experimental): Stage 1: Support, facilitate, and assist in linkage to PrEP clinic and to facilitate initiation of, and obtaining, PrEP medications.
  Interventions: Behavioral: PrEPare for Work: Strength Based Case Management (Stage 1)
- PrEP adherence training and counseling (Experimental): Stage 2: Up to three adherence training and counseling intervention sessions (once per week for two to three weeks) with a clinical interventionist.
  Interventions: Behavioral: PrEPare for Work: Adherence Training and Counseling (Stage 2)
- Standard of Care:Stage 1 (No Intervention): Stage 1: Referral to The Miriam Hospital PrEP Clinic.
- Standard of Care: Stage 2 (No Intervention): Stage 2: Doctor visit every three months to assess for side effects and receive a HIV test.

INTERVENTIONS:
Behavioral: PrEPare for Work: Strength Based Case Management (Stage 1) — Support, facilitate, and assist in linkage to PrEP clinic and to facilitate initiation of, and obtaining, PrEP medications.
  Arms: Strength Based Case Management
Behavioral: PrEPare for Work: Adherence Training and Counseling (Stage 2) — Up to three adherence training and counseling intervention sessions (once per week for two to three weeks) with a clinical interventionist.
  Arms: PrEP adherence training and counseling

SUMMARY:
"PrEPare for Work" is a two-stage randomized controlled pilot trial which utilizes a behavioral intervention to optimize the uptake and adherence of Pre-exposure Prophylaxis (PrEP) in Male Sex Workers (MSW).

DETAILED DESCRIPTION:
The "PrEPare for Work" package includes two behavioral intervention components:

1. Strengths-based case management for PrEP initiation, and
2. Counseling and problem-solving PrEP adherence intervention that addresses individualized barriers to optimal use.

Stage 1: MSW will be equally randomized to receive either the strengths-based case management or standard of care referral to PrEP clinic.

Stage 2: Those from stage 1 who initiate PrEP , regardless of stage 1 randomization condition, will then be equally randomized to either the "PrEPare for Work" adherence intervention or standard of care comparison condition.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Biological male at birth and current male gender identity
* Exchanged sex for money or drugs with another man in the past 3 months
* Report behavioral risk for HIV infection, consistent with Centers for Disease Control and Prevention guidelines for prescribing PrEP: condomless anal intercourse with at least one HIV-infected or unknown serostatus partner in the past three months
* HIV uninfected by antibody test* Stage 2
* Able to understand and speak English (for consent and counseling)
* Mental competency to provide voluntary informed consent
* Lives in the New England area
* Willing to initiate PrEP

Exclusion Criteria:

* Unable to provide informed consent, including as a result of severe mental illness requiring immediate treatment or mental illness limiting the ability to participate
* HIV Positive at baseline
* Infected with Hepatitis B or diagnosed with renal insufficiency (glomerular filtration rate < 50) *Stage 2
* History of or current medical conditions that would preclude taking Truvada for PrEP *Stage 2
* Currently taking Truvada for PrEP

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological male at birth and current male gender identity
Enrollment: 111 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Mimiaga, ScD, MPH, Principal Investigator — Brown University, School of Public Health, Center for Health Equity Research
Locations (2):
- United States (2):
  - The Miriam Hospital, Providence, Rhode Island
  - Brown University School of Public Health, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated that this data will be presented annually on data collected after the second year when sufficient baseline data is collected. It is anticipated that most of the papers and data-based projects/presentations will happen in year 3, when all of the baseline data is collected, and the 3 month outcome has occurred for all participants. Sharing of the findings will involve a primary paper describing the study outcome and a paper that describes the intervention, as well as submitting to lead workshops on the intervention approach at relevant national meetings and conferences. Raw data for additional analysis will be available to outside individuals through contacting the MPIs. Information regarding the availability of data for analysis will be listed on the MPIs' web pages. Contact information for the MPIs will be listed in all manuscripts and publications as another means to access data.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was partially enrolled and never completed enrollment. Only participants who completed Stage 1 AND who initiated PrEP were included in Stage 2.
Period: Stage 1: PrEP Uptake
Arm/Group | Strength Based Case Management | Standard of Care:Stage 1 | PrEP Adherence Training and Counseling | Standard of Care: Stage 2
Started | 55 | 55 | 0 (This intervention was not provided until Stage 2) | 0 (This intervention was not provided until Stage 2)
Completed | 44 | 45 | 0 | 0
Not Completed | 11 | 10 | 0 | 0
Not completed — Incarcerated | 3 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 0 | 0
Not completed — Lost to Follow-up | 6 | 5 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Period: Stage 2: PrEP Adherence
Arm/Group | Strength Based Case Management | Standard of Care:Stage 1 | PrEP Adherence Training and Counseling | Standard of Care: Stage 2
Started | 0 (This was only provided in Stage 1) | 0 (This was only provided in Stage 1) | 17 (Only individuals who completed Stage 1 AND initiated PrEP were randomized in Stage 2.) | 18 (Only individuals who completed Stage 1 AND initiated PrEP were randomized in Stage 2.)
Completed | 0 | 0 | 11 | 16
Not Completed | 0 | 0 | 6 | 2
Not completed — Incarcerated | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Population: This was a two-stage sequential randomization design. Therefore, all of those in the Stage 2 arms (PrEP adherence training and counseling and Standard of Care) are already counted in Stage 1 arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Strength Based Case Management | Standard of Care:Stage 1 | PrEP Adherence Training and Counseling | Standard of Care: Stage 2 | Total
Number analyzed (Participants) | 55 | 55 | 0 | 0 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (7.8) | 34.6 (9.2) |  |  | 34.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 |  |  | 0
  Male | 55 | 55 |  |  | 110
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 27 | 35 |  |  | 62
  Black, non-Hispanic | 8 | 7 |  |  | 15
  Hispanic/Latino | 15 | 9 |  |  | 24
  Other | 5 | 4 |  |  | 9
Region of Enrollment [Number; unit: participants]
  United States | 55 | 55 |  |  | 110
PrEP Use Self-Efficacy [Mean (Standard Deviation); unit: units on a scale] — Summary measure - range 0-10, with higher scores indicating higher self-efficacy for using PrEP
  units on a scale | 7.1 (3.2) | 7.7 (2.1) |  |  | 7.4 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Verified Attendance at Initial Appointment at PrEP Clinic
Description: Number of participants with attendance at initial appointment at PrEP Clinic verified using medical records
Time Frame: 2-month post Stage 1 randomization
Population: Per study design, linkage to PrEP care was only assessed in Stage 1; Additionally, because this was based on medical records we could include anyone that was not withdrawn or incarcerated or had died (n=5 in each arm).
Measure: Count of Participants; unit: Participants
Arm/Group | Strength Based Case Management | Standard of Care:Stage 1
Number analyzed (Participants) | 50 | 50
Participants | 30 | 13

2. Primary Outcome: Number of Participants Who Initiated PrEP
Description: Initial prescription from provider filled and shown to study staff
Time Frame: 2-month post Stage 1 randomization
Population: Per study design, PrEP initiation was only assessed in Stage 1; Additionally, because this required proof of prescription, we excluded those who were loss to follow up for Stage 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Strength Based Case Management | Standard of Care:Stage 1
Number analyzed (Participants) | 44 | 45
Participants | 26 | 9

3. Primary Outcome: Number of Participants Reporting Optimal PrEP Adherence
Description: Self-reporting missing 0 PrEP pills in the past week
Time Frame: 6-months post Stage 2 randomization
Population: Per study design, PrEP adherence was only assessed in Stage 2 (and among Stage 2 participants); Additionally, because this was based on self-report, PrEP adherence was only assessed among those with follow up data.
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP Adherence Training and Counseling | Standard of Care: Stage 2
Number analyzed (Participants) | 11 | 16
Participants | 5 | 5

ADVERSE EVENTS:
Time Frame: For participants only in Stage 1, adverse event data were collected for approximately 2 months for each participant. For participants subsequently randomized into Stage 2, adverse event data were collected for an additional 6 months for each participant.
Arm/Group | Strength Based Case Management | Standard of Care:Stage 1 | PrEP Adherence Training and Counseling | Standard of Care: Stage 2
All-Cause Mortality (participants affected / at risk) | 1/55 | 2/55 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 3/17 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strength Based Case Management (N=55) | Standard of Care:Stage 1 (N=55) | PrEP Adherence Training and Counseling (N=17) | Standard of Care: Stage 2 (N=18)
Potential Disclosure (Social circumstances) | 0 | 0 | 1 (1) | 0
Homicidal ideation (Social circumstances) | 0 | 0 | 1 (1) | 0
Police involvement (Social circumstances) | 0 | 0 | 1 (2) | 0 — Using study phone to call police (but then hang up)

LIMITATIONS AND CAVEATS:
Due to COVID, we are delayed in receiving the results of our biomarkers (specifically, hair analysis for PrEP adherence).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT03086057/ICF_000.pdf
  • Study Protocol (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT03086057/Prot_001.pdf
  • Statistical Analysis Plan (2015-09-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT03086057/SAP_002.pdf